CLINICAL TRIAL: NCT06501820
Title: Neural Control of Gait & Navigation in ADRD, Aim 3 Clinical Trial
Brief Title: Neural Control of Gait & Navigation in ADRD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB202400767; R01AG089050 (NIH)
Record Dates: First submitted 2024-06-24; First posted 2024-07-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Aging
Keywords: aging; subjective cognitive decline; vestibular; mobility
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Two group, repeated measures, double blind active or sham stimulation
Who Masked: Participant, Investigator
Masking Description: Sham transcranial magnetic stimulation is extremely effective. It involves current ramp up and down, resulting in potential tingling of the scalp similar to active stimulation. The investigator will also be blinded; they will enter a code into the stimulation box that results in either active or sham stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sham stimulation (Sham Comparator): The tDCS electrodes are applied and the current ramps up and then down, resulting in a very effective sham condition.
  Interventions: Device: Transcranial direct current stimulation
- Active stimulation (Experimental): Transcranial direct current stimulation, bilateral, 2 mA, applied to the vestibular cortex.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — 2mA transcranial direct current stimulation, applied bilaterally on the scalp, over the brain vestibular cortex

SUMMARY:
Brain network segregation, or independent functioning, declines with age and is associated with slower walking speed. Here, the investigators will determine the extent to which brain vestibular network segregation can be altered with bilateral vestibular cortical transcranial direct current stimulation (tDCS) in older adults with subjective cognitive decline. Participants will be randomly assigned to an active or sham stimulation condition. They will receive three, 20-minute sessions of tDCS while they are walking and performing cognitive tasks. MRI of the brain will be acquired before and after these three sessions.

DETAILED DESCRIPTION:
The investigators will conduct this experiment with individuals that have subjective cognitive decline. At pre- and post-test, they will receive structural MRI and resting state fMRI so that we can quantify brain vestibular-motor and vestibular-hippocampal network segregation. These will serve as the primary outcome metrics.

Participants will perform a walking + spatial navigation task. Their performance in the first 15 minutes will count as their pre-test behavioral score (gait speed, gait variability, navigation path integration task error). Participants will then receive either sham or active bilateral vestibular cortical tDCS. They will be randomly assigned into the active (n=30) or sham tDCS group (n=30) without their awareness. The active group will receive 20 minutes of 2mA tDCS bilaterally to the vestibular cortex (right parietal operculum 2 (OP2), MNI coordinates 50,-32,18; left OP2, MNI coordinates 38,-20,16); these regions have been identified through meta-analyses as being responsive to various types of vestibular stimulation. Electrodes will be placed using a Brainsight (Rogue Research, Montreal, QC, Canada) neuro-navigation system in which we will fit each participant's head to a standardized template space (MNI 152 template) from their MRIs (neuro-navigated stimulation). The anode electrode will be placed over the left vestibular cortex, whereas the cathode will be placed over the right. Stimulation at 2 mA has previously been shown to result in net excitation in both regions stimulated, as opposed to the traditional approach that increases excitability under the anode and inhibits excitability under the cathode. The sham tDCS group will receive stimulation for only 30 seconds during an active ramp up, and then immediate ramp down. This is to ensure that neither group is actively aware if they are receiving tDCS stimulation. The experimenter will also be blinded to whether a participant is receiving active or sham stimulation; they will enter a code into the stimulation box, making the protocol double blind. Participants will perform walking + spatial navigation on three days for 30 minutes per day (tDCS will be on for the first 20 minutes), under either active or sham stimulation. This protocol will be applied over three sessions, each separated by at least 24 hours and all three completed within 10 days.

The investigators will determine whether bilateral tDCS increases vestibular-motor and vestibular-hippocampal network segregation. They will examine behavioral task improvements as secondary outcomes. Using an ANOVA model, a total sample size of 60 (n=30 per group) results in 80% power to detect an effect size as small as Cohen f= 0.37 at significance level 0.05. Using a two-sided two-sample t-test with the same sample size, power and significance level (if the investigators were to analyze each variable separately), the minimum detectable effect size is 0.75 and for a nonparametric Wilcoxon-Mann-Whitney test, it becomes 0.76 under the same settings.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling men and women 18-35 years old or 65-89 years old
* Ability to walk unassisted for ten minutes
* Willingness to undergo all testing procedures
* English speaking Additional Inclusion Criteria for those with SCD
* Subjective report of cognitive complaints with scores >16 on the Cognitive Change Index (CCI-20), a validated scale of subjective cognitive decline (Saykin et al., 2013). This scale consists of 20 items that are rated on 5 point Likert scale, where 1= "Normal: No change compared to 5 years ago", 3= "Mild Problem: Some change compared to 5 years ago) and 5="Severe Problem: Much worse compared to 5 years ago".)
* No evidence of dementia or mild cognitive impairment based on cognitive screening (i.e., Montreal Cognitive Assessment (MoCA) score within normal limits for age, education and sex using the NACC Uniform Data Set (UDS) norms (Weintraub et al., 2018)[119]
* No psychometric evidence of cognitive impairment based on performance on the Neuropsychological Battery from the NACC Unified Data Set, version 3[119]. The battery includes measures of attention, recent memory, language, visuospatial, and executive function. Norms are available for over 3600 older adults [119]. Scores on these measures cannot be lower than 1.0 SD (16th %ile) below normative values based on age, education, and gender.
* Reading at > 8th grade level based on the reading subtest of the Wide Range Achievement Test- IV.
* Global Clinic Dementia Rating (CDR) score must be 0 [156]
* Family history of dementia/probable Alzheimer's disease in first degree relative (parents, children, siblings)
* Normal functional behavior in terms of daily activities, based on the Functional Activities Scale[122]
* In line with recommendations of SCD task force (Molienueva et al., 2017)[116] an informant must be available for two reasons: a) to provide information about the participant's complaints using the informant version of the CCI-20, and b) to corroborate normal IADL's on the Functional Activity Questionnaire[120] .

Exclusion Criteria:

* Significant medical event requiring hospitalization in the past 6 months that has the potential to contaminate data being collected (fracture, hospitalization etc.)
* Severe visual impairment or corrected visual acuity less than 20/40, which would preclude completion of the assessments
* Inability to undergo brain imaging due to claustrophobia or implants such as pacemakers, heart valves, brain aneurysm clips, orthodontics, non-removable body jewelry, or shrapnel containing ferromagnetic metal
* tDCS ineligibility for Aim 3 (history of epilepsy, medications that alter cortical excitability, etc.)
* History of stroke
* Any history of clinically diagnosed traumatic brain injury resulting in > 1 minute loss of consciousness
* Any major ADL disability (unable to feed, dress, bath, use the toilet, or transfer)
* Report of lower extremity pain due to osteoarthritis that significantly limits mobility
* Diagnosis or treatment for rheumatoid arthritis
* Known neuromuscular disorder or overt neurological disease (e.g. Multiple Sclerosis, Rhabdomyolysis, Myasthenia Gravis, Ataxia, Apraxia, post-polio syndrome, mitochondrial myopathy, Parkinson's Disease, ALS etc.)
* Unable to communicate because of severe hearing loss or speech disorder
* Planned surgical procedure or hospitalization in the next 12 months (joint replacement, coronary artery bypass graft, etc.)
* Severe pulmonary disease, requiring the use of supplemental oxygen
* Terminal illness, as determined by a physician
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, recent history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Is planning to move out of the area during the follow up period
* Use of walker or wheel chair
* Failure to provide informed consent

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Vestibular network segregation score, measured with functional MRI | Pre-intervention, within 1 week post-intervention
  Independence of brain network functioning

SECONDARY OUTCOMES:
Gait variability, measured with an inertial measurement unit on the sacrum | Intervention is applied while participants are walking
  Variability of walking
Path integration error, measured in degrees | Intervention is applied while this task is performed
  Navigation task performance

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Seidler, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified brain and behavioral data will be shared via Open Science Framework and other databases.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Following completion of the study and publication of results, the data will be available indefinitely.
Access Criteria: Data will be accessible